CLINICAL TRIAL: NCT04509115
Title: Real-World Data to Assess Variation in Opioid Prescribing and Use for Acute Pain in Diverse Populations
Brief Title: Variation in Opioid Prescribing and Use for Acute Pain in Diverse Populations
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2000027561; 2U01FD005938-03 (FDA)
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Opioid Use; Opioid Prescribing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients given short-acting opioid prescription: Patients not currently using opioids who receive a new short-acting opioid prescription for acute pain will be recruited.
  Interventions: Drug: Short-acting opioid prescription for acute pain

INTERVENTIONS:
Drug: Short-acting opioid prescription for acute pain — Patients not currently using opioids who receive a new short-acting opioid prescription as part of routine care for acute pain will be recruited and followed prospectively for 180 days.

SUMMARY:
This study will characterize patient pain and opioid use after an initial opioid prescription for acute pain.

DETAILED DESCRIPTION:
The purpose of this study is to characterize patient pain and opioid use after an initial opioid prescription for acute pain. The investigators aim to enroll a total of 300 patients receiving a prescription for an opioid in primary and urgent care, inpatient care (child birth and total knee arthroplasty), and in the emergency department. Patients not currently using opioids who receive a new short-acting opioid prescription for acute pain will be recruited and followed prospectively for 180 days to assess pain trajectories, analgesic and non-pharmacologic treatment use, activity, and health care service use. The patient-centered health data sharing platform (Hugo) will be used to collect patient-reported outcomes and structured data from pharmacy and electronic health records patient portals as well as patient-generated data collected through personal digital devices (Fitbit).

Specific aims

1. To assess patients' pain and opioid use patterns in episodes of acute pain for which opioids were prescribed, characterizing pain severity and persistence, as well as other prescription and over-the-counter pain medication use
2. To examine associations between patient demographic, clinical and emotional characteristics and outcomes of pain severity and persistence, opioid and non-opioid treatment patterns, satisfaction with care, and barriers to care
3. To assess how patients handled unused opioids

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* Experiencing acute pain of less than 8 weeks duration at the time the opioid is prescribed
* Received prescription for opioid analgesic at visit; opioids included in the study will be all FDA-approved enteral, transdermal, and transmucosal opioid analgesics including the most common: hydrocodone (except cough and anti-diarrheal medications), oxycodone, codeine (except cough medications), tramadol, morphine, hydromorphone. Receipt of a prescription for the following is not an exclusion: buprenorphine (as an analgesic), butorphanol, dihydrocodeine, fentanyl, meperidine, methadone (as an analgesic), oxymorphone, pentazocine, sufentanil, and tapentadol. All of these opioids are included in any combinations with acetaminophen, aspirin, ibuprofen, naloxone, etc.
* Self-report of no opioid use (no use of prescribed opioids or illicit opioids, including medical or non-medical use) in the past 6 months
* Willing and able to give consent and participate in study
* Able to access a device with web access (laptop, desktop, smartphone, or tablet) daily to complete study surveys
* Willing to connect Fitbit to a mobile device (smartphone or tablet) that can regularly link to Hugo for data transfer
* Willing to use the health data sharing platform
* Released/discharged to home after their visit.

Exclusion Criteria:

* Pain thought to be caused by a systemic disease very likely to progress to chronic pain (e.g., sickle cell disease, fibromyalgia, lupus, multiple sclerosis, etc.);
* Cancer or end-of-life pain;
* Unable to give consent and be enrolled within 3 days of their visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit a total of 1,550 patients receiving primary and urgent care, emergency department care, inpatient care (child birth and total knee arthroplasty), and dental care in 5 healthcare systems. Participants must be 18 years or older, be English- or Spanish-speaking, and be willing and able to consent for themselves.
Sampling Method: Non-Probability Sample
Enrollment: 1709 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Opioid Pain medication use | From baseline up to 180 days
  Number of days using any opioid medications
Non-Opioid pain medication and treatment use | From baseline up to 180 days
  Number of days using any non-opioid drugs/treatments
Pain medication use concordant with directions for use | From baseline up to 180 days
  Comparison of directions for use and actual use: For each day the person takes opioids, measure whether the number of pills taken falls within the range prescribed, below the prescribed range, or above the prescribed range. The overall proportion of days taking less than the prescribed range, within the prescribed range, and over the prescribed range will be calculated for each patient and the distribution of these measures will be plotted as histograms and reported as the median, 25th percentile and 75th percentile.

SECONDARY OUTCOMES:
Time to opioid discontinuation | From initial opioid use to the day on which the last opioid was taken, up to 180 days.
  Discontinuation defined as 30 days with no opioid use. . If 30 days pass with no opioid use, but the participant takes an opioid on the 31st day, a new episode of opioid use will be considered to have started and the time to opioid discontinuation will again be measured.
Time to pain resolution | From baseline up to 180 days
  Pain resolution will be defined as patient no longer indicating pain in the body area initially treated, as indicated by either a) an overall pain rating of 0 on the brief pain inventory scale from 0 to 10, with 0 being no pain and 10 the worst pain imaginable, or b) the patient no longer selects the body area initially treated when completing the body map of areas where patient is experiencing pain).
Average activity levels | From baseline up to 180 days
  Trajectory of the average steps per day registered by the Fitbit Inspire over time (decreasing, increasing, stable) for the periods between enrollment and stopping opioids, enrollment and pain resolution
Treatment satisfaction | From baseline up to 180 days
  Patient-reported satisfaction with health care received to treat pain: distribution of responses. "Treatment satisfaction: In general, how satisfied are you with the health care you received to treat your pain? Very satisfied; Somewhat satisfied; Somewhat dissatisfied; Very dissatisfied"
Barriers to treatment | From baseline up to 180 days
  Reported barriers to accessing additional treatment: proportion reporting difficulty with one or more of the following: getting a refill, difficulty getting a pharmacy to fill, getting insurance to pay for treatment, being able to afford to pay for treatment.
Description of pain medications used | From baseline up to 180 days
  Use patterns of different pain medications (opioid and any combination ingredients), including the strength, and number of pills dispensed (in MME)
Patient opioid use progression | From baseline up to 180 days
  Proportion of patients progressing to: long-term use of opioids (90+ days of use or 120+ days' supply filled)
Patient chronic pain progression | From baseline up to 180 days
  Proportion of patients progressing to chronic pain (pain lasts 90+ days)
Patient-Reported Outcomes Measurement Information System (PROMIS) Prescription Pain Medication Misuse short-form; selected items | From baseline up to 180 days
  We will assess this outcome with 5 survey items drawn from the Patient-Reported Outcomes Measurement Information System (PROMIS) Prescription Pain Medication Misuse short-form. The total score for these 5 items ranges from 5 to 25 with 25 signaling greatest misuse.
Storage and disposal guidance | From baseline up to 180 days
  Proportion of patients that report receiving: information on how to properly dispose of medication, and/or on the importance of disposing of unused medication.
Opioid Storage Methods | From baseline up to 180 days
  Proportion of patients that report storing opioids in: a locked location (proportion reporting always or almost always), a latched location (proportion reporting always or almost always), in the original bottle (proportion reporting always or almost always)
Unused Opioids | From baseline up to 180 days
  Number of opioids left over after opioid discontinuation and estimated amount used during study period Measured in absolute amounts-e.g., mg of oxycodone-as well as MME and tablets
Estimated Opioid Use | From baseline up to 180 days
  Based on left over opioids, amount used during study period Measured in absolute amounts-e.g., mg of oxycodone-as well as MME and tablets
Opioid Disposal | From baseline up to 180 days
  Proportion of patients reporting each disposal method including disposing of drug in garbage, flushed down toilet, returned to police, returned to pharmacy, passed on to someone else, kept for future use/did not dispose, used up all opioids. Motivations for disposing of or keeping leftover drugs, proportion reporting each survey response.
Motivations for disposing or keeping leftover drugs | From baseline up to 180 days
  We will assess this outcome with 16 survey items drawn from the University of South Florida and Purdue Pharma study of disposal. We will report on the proportion of participants endorsing each item. Representative items include inconvenience, risk of disposal, and potential need for opioids in the future

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ross, MD, MHS, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Cedars Sinai, Los Angeles, California
  - Yale-New Haven Health, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota
  - Monument Health, Rapid City, South Dakota

REFERENCES:
- [Derived] Jeffery MM, Ahadpour M, Allen S, Araojo R, Bellolio F, Chang N, Ciaccio L, Emanuel L, Fillmore J, Gilbert GH, Koussis P, Lee C, Lipkind H, Mallama C, Meyer T, Moncur M, Nuckols T, Pacanowski MA, Page DB, Papadopoulos E, Ritchie JD, Ross JS, Shah ND, Soukup M, St Clair CO, Tamang S, Torbati S, Wallace DW, Zhao Y, Heckmann R. Acute pain pathways: protocol for a prospective cohort study. BMJ Open. 2022 Jul 5;12(7):e058782. doi: 10.1136/bmjopen-2021-058782. PMID 35790333